CLINICAL TRIAL: NCT06286748
Title: Effects of Beetroot Extract Supplementation Associated With an Exercise Protocol on Oxidative Stress, Inflammation, and Functional Capacity in Patients With Chronic Kidney Disease
Brief Title: Beetroot Extract Supplementation Associated With an Exercise Protocol for Chronic Kidney Disease Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal Fluminense (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: DeniseMafra19
Record Dates: First submitted 2024-02-11; First posted 2024-02-29 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Chronic Kidney Diseases
Keywords: chronic kidney disease; beetroot; exercise; inflammation; oxidative stress
MeSH Terms: conditions — Renal Insufficiency, Chronic; Motor Activity; Inflammation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): Beetroot juice + exercise. Patients will ingest 200ml of beet juice (Beta vulgaris) containing approximately 300mg of nitrate (NO3-), and after 2 hours they will be instructed to perform an exercise protocol.
  Interventions: Dietary Supplement: Beetroot juice
- Placebo (Placebo Comparator): Placebo + exercise. Patients will ingest 200ml of placebo (water, without nitrate (NO3-)), and after 2 hours they will be instructed to perform an exercise protocol.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Beetroot juice — Beetroot juice + exercise. Patients will ingest 200ml of beet juice (Beta vulgaris) containing approximately 300mg of nitrate (NO3-), and after 2 hours they will be instructed to perform an exercise protocol.
  Arms: Intervention
Other: Placebo — Placebo + exercise. Patients will ingest 200ml of placebo (water, without nitrate (NO3-)), and after 2 hours they will be instructed to perform an exercise protocol.
  Arms: Placebo

SUMMARY:
Chronic kidney disease (CKD) patients often present systemic inflammation and oxidative stress, resulting in metabolic disorders and high rates of disease-associated cardiovascular death. The literature has indicated that dietary control, the use of bioactive compounds, and the practice of regular physical exercise are essential for the prevention and management of CKD and its complications. In this context, beetroot (Beta vulgaris rubra) deserves attention as it is a source of several bioactive compounds, such as nitrate, betaine, and betalain, with beneficial effects for CKD patients, including anti-inflammatory, antioxidant effects, reduction of blood pressure, and vasodilatory action. The antioxidant and anti-inflammatory properties, in addition to their vasodilatory and antihypertensive capacity, can make supplementation of beetroot an excellent nutritional strategy to help in the treatment of CKD patients. So, this research project will bring contributions to the scientific world, providing strategies for application in clinical practice and the care of patients with CKD, on the use of beetroot associated with an exercise protocol as a non-pharmacological strategy in modulating inflammation, oxidative stress, and improved functional capacity. Furthermore, when supplemented hours before physical training, has been identified as an important factor in improving performance in these activities. Therefore, this study aims to evaluate the effects of supplementation (acute and chronic) of beetroot extract associated with an exercise protocol on complications associated with CKD.

DETAILED DESCRIPTION:
This is an acute and chronic study, the acute type being a randomized, double-blind, crossover clinical trial with a washout period and placebo-controlled trial (RCT), and the chronic concerns a randomized, double-blind, placebo-controlled clinical trial type study (randomized controlled trial - RCT). To calculate the sample size, it was assumed that the tumor necrosis factor (TNF)-alpha concentration would decrease by 1.0 pg/mL after intervention with beetroot juice using the within-patient standard deviation of 2.3. It was assumed a type I error of P < 0.05 and a test power of 80%, and it was estimated that, for both the acute and chronic study, 25 patients would be needed (margin of 10%, 28 patients) with CKD undergoing conservative treatment at the Renal Nutrition Outpatient Clinic. Eligible patients of both genders, previously evaluated and authorized by the medical and nutritionist staff, will be invited to participate in the research in person and verbally, during nutritional consultations at the Renal Nutrition Outpatient Clinic. The acute intervention study will be divided into 3 stages. The first stage will consist of collecting anthropometric data, food intake, completion of individual quality of life questionnaires (SF-36) and physical activity level (IPAQ) and, finally, familiarization with the exercise protocol that will be carried out in the following stages. Already in second stage, initial data will be collected from participants, soon after, participantes will be invited to perform the 6-minute walk test. Then, all individuals will be instructed to ingest beetroot juice or placebo and wait for at least 2 hours. After 2 hours, all volunteers must complete the training protocol lasting 20 minutes. At the end of the exercises, both groups will be reevaluated. Finally, in the third and final stage, after 14 washout days participants will go through the same process described in the previous stage, however, participantes will carry out the opposite intervention to that carried out in stage two, that is, those who participated in the beetroot juice group will become part of the control group and vice versa. The chronic intervention study will be similar to the acute intervention stages, but individuals will undergo three weekly sessions, totaling 24 training sessions (8 weeks), without washout period. The second stage will begin with the collection of blood samples and vital data of participants, as well as the performance. For eight weeks, volunteers will ingest beetroot juice or control and, after 2 hours of rest, they must perform the protocol of circuit exercises. The end of this stage will be characterized by the collection of blood, vital signs, data on food intake, clinical, anthropometric, filling out questionnaires (SF-36 and IPAC) and carrying out. Before and after training, each practitioner's vital signs will be measured by security measure. If the resting heart rate is greater than 120 beats per minute (bpm), systolic blood pressure greater than 180 mmHg or diastolic blood pressure greater than 100 mmHg, the patient will be contraindicated to perform the day's training. Training should also be stopped if the subject presents chest pain, dyspnea, lower leg cramps, staggering gait, intense sweating and paleness, recommendations that will also be adopted to perform.

ELIGIBILITY:
Inclusion Criteria:

* Patients with CKD undergoing conservative treatment (stages G3a-G4);
* Aged between 18 and 65 years old;
* Patients undergoing nutritional monitoring for more than 6 months.

Exclusion Criteria:

* Patients using catabolic drugs;
* Smokers
* Pregnant women;
* Using antibiotics and of proton pump inhibitors in the last 3 months;
* Antioxidant supplements and habitual intake of beetroot or nitrate supplement;
* Those who are clinically unstable (unstable angina, atrial fibrillation, significant cardiac arrhythmia and acute illness in the last month; and glycemic lability);
* Unable to exercise (amputation without prosthesis); musculoskeletal pain at rest or with minimal physical activity, inability to sit or walk without assistance, use of a walking device, dyspnea at rest or with light exertion;
* Those with autoimmune diseases and infectious diseases, cancer, liver disease and AIDS.
* Patients with parathormone (PTH) levels above 500pg/mL;
* Those who are allergic or intolerant to the components of the juice.
* Patients with any impediment to completing the proposed exercise protocol, such as due to travel or difficulty accessing the location where the research will be carried out.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-04-10 (Actual); Primary Completion 2025-12-10 (Estimated); Study Completion 2026-12-10 (Estimated)

PRIMARY OUTCOMES:
Change individual quality of life | 8 weeks
  Qualitative parameter
Change physical activity level | 8 weeks
  Qualitative parameter

CONTACTS AND LOCATIONS:
Overall Officials: Denise Mafra, PhD, Principal Investigator — Associate Professor - Universidade Federal Fluminense
Locations (1):
- Denise Mafra, Rio de Janeiro, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No